CLINICAL TRIAL: NCT04971616
Title: Risk Screening and Assessment of Shoulder, Neck and Lower Back Discomfort.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020342
Record Dates: First submitted 2021-06-27; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Low Back Pain; Neck Pain; Shoulder Pain
MeSH Terms: conditions — Low Back Pain; Neck Pain; Shoulder Pain | interventions — Demography; Range of Motion, Articular

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with shoulder, neck and lower back discomfort: Patients with shoulder, neck and lower back discomfort.
  Interventions: Other: Demographic data and range of motion.

INTERVENTIONS:
Other: Demographic data and range of motion. — The body parameters (BMI, age, gender), daily activities (daily steps, sedentary), work and rest time (sleep time, quality) were collected through wearable devices. The range of motion of neck and waist was collected through hand-held devices.

SUMMARY:
Identifying high-risk factors that may lead to shoulder, neck and lower back discomfort and contributing to the primary prevention of disease progression.

DETAILED DESCRIPTION:
The purpose of this study is to design a self-assessment scheme for clinical assessment of shoulder, neck and lower back function and compare the consistency between clinical assessment and self-assessment. The body parameters (BMI, age, gender), daily activities (daily steps, sedentary), work and rest time (sleep time, quality) were collected through wearable devices, evaluating the risk factors of shoulder, neck and lower back discomfort.

ELIGIBILITY:
Inclusion Criteria

* 20-40 year of age with symptoms of shoulder
* Neck and lower back discomfort

Exclusion Criteria

* Red flag sign of the neck

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20-40 year of age with shoulder, neck and lower back discomfort
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Range of motion (ROM) of the neck | at least 2-week monitoring by wearable devices
  Patients' range of motion of the neck in all directions are measured using hand-held devices.
Oswestry Disability Index (ODI) | at least 2-week monitoring by wearable devices
  Oswestry Disability Index of the neck is collected for the evaluation of neck functions.
Visual Analogue Scale (VAS) | at least 2-week monitoring by wearable devices
  Visual Analogue Scale is collected for pain assessment.
Roland-Morris Disability Questionnaire (RDQ) | at least 2-week monitoring by wearable devices
  Roland-Morris Disability Questionnaire is collected for the evaluation of lower back functions.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-quan Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No